CLINICAL TRIAL: NCT04408469
Title: A Randomized Controlled Trial of Online LGBTQ-affirmative Cognitive Behavioral Therapy to Reduce Depression and Associated Health Risks Among Young Adults
Brief Title: A Trial of Online LGBTQ-affirmative Cognitive Behavioral Therapy to Reduce Depression and Associated Health Risks Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2000025803
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-11

CONDITIONS: LGBTQ; Sexual Behavior
Keywords: on-line intervention
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online EQuIP (Experimental): The online CBT treatment consists of 10 weekly modules that participants will complete over the course of 10 weeks.
  Interventions: Behavioral: Online EQuIP
- Self-Monitoring (Placebo Comparator): Participants will be asked to indicate their past 7-day mood; stress experiences; and mental and behavioral health on an online survey experience once per week for 10 weeks
  Interventions: Behavioral: Self-monitoring control

INTERVENTIONS:
Behavioral: Online EQuIP — This online CBT treatment consists of 10 weekly modules that participants will complete over the course of 10 weeks.
  Arms: Online EQuIP
Behavioral: Self-monitoring control — Participants will be asked to indicate their past 7-day mood; stress experiences; and mental and behavioral health on an online survey experience once per week for 10 weeks
  Arms: Self-Monitoring

SUMMARY:
This study is to test the efficacy of an online CBT intervention (EQuIP) that addresses the pathways through which minority stress compromises LGBTQ young adults' co-occurring mental (e.g., depression) and behavioral (e.g., substance use, condomless anal sex) health problems. This purpose of this study is to determine if the treatment is efficacious when delivered online and if its efficacy exceeds that of the self-monitoring control.

DETAILED DESCRIPTION:
To evaluate the preliminary efficacy of an LGBTQ-affirmative online CBT treatment and whether such an LGBTQ-affirmative focus adds benefit, a 2-arm RCT that would examine (1) whether online EQuIP demonstrates significant mental health improvements compared to self-monitoring of stress and mood, and (2) whether participant baseline LGBTQ-specific stress exposure moderates treatment efficacy, such that participants with the most LGBTQ-specific stress exposure benefit more from online EQuIP than self-monitoring of stress and mood.

The primary outcomes are depressive symptoms, anxiety symptoms, substance abuse, sexual risk behavior, and suicidality, all of which disproportionally affect LGBTQ young adults. Secondary outcomes include hypothesized cognitive, affective, and behavioral minority stress mechanisms, such as internalized homophobia, rejection sensitivity, concealment, social isolation, and emotional dysregulation.

Participants will be randomized to either self-monitoring control or Online EQuIP group.

Self-monitoring control: In this control condition, participants will be asked to indicate their past 7-day mood; stress experiences; and mental and behavioral health on an online survey. This type of self-monitoring has been shown to yield improvement in behavioral health outcomes. Self-reporting LGBTQ stress experiences has also been shown to produce reductions in depression symptoms over time. Participants will record these experiences once per week for 10 weeks.

Online EQuIP: This online CBT treatment consists of 10 weekly modules that participants will complete over the course of 10 weeks. Modules contain weekly psychoeducational text and vignettes about minority stress and mental health; brief videos illustrating the CBT skills; and homework exercises that therapists review and provide feedback on. Homework exercises include weekly tracking of stressful situations and mood, practicing new skills (e.g., mindfulness, cognitive restructuring), and exercises related to considering the origins of stress and negative emotions that participants may be experiencing. Therapists provide feedback after each homework assignment, including reviewing each participant's treatment goals as part of the first session's homework. Therapists who support this condition will be instructed to incorporate LGBTQ-specific content and feedback into homework reviews. Therapists will either be postdoctoral fellows in the Pachankis lab or clinical/counseling psychology interns/externs in the Pachankis lab who possess an advanced degree in a mental health field with significant prior experience treating LGBTQ young adults with mental health concerns. Modules were adapted directly from the in-person materials (e.g., therapist manual, participant handouts) used in our previously successful trials of this treatment. A team of six therapists and supervisors of the original in-person treatment adapted the text for the online modules, including realistic vignettes and easy-to-follow skills training. A video production company created accompanying videos with our clinical team's close input.

In preparation for this RCT, the online EQuIP treatment was delivered to 14 LGBTQ young adults who meet all eligibility criteria for the full trial. The purpose of this initial test was to ensure acceptability of the treatment content and usability of the technical platform.

ELIGIBILITY:
Inclusion Criteria:

* identify as lesbian, bisexual, gay, or another sexual minority identity (e.g., pansexual, demisexual)
* past-week symptoms of depression or anxiety using the Brief Symptom Inventory-4 cutoff of 2.5 on either the depression subscale or anxiety subscale
* weekly access to internet on a laptop, desktop, or tablet device
* ability to read, write, and speak in English
* provision of informed consent.

Exclusion Criteria:

* current active suicidality or homicidality (defined as active intent or concrete plan, as opposed to passive suicidal ideation)
* evidence of active untreated mania, psychosis, or gross cognitive impairment - current enrollment in an intervention study
* current enrollment in intensive mental health treatment (i.e., receiving mental health treatment more than once per month or 8 or more sessions of CBT within the past year.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participant identifies as lesbian, bisexual, gay, or another sexual minority identity (e.g., pansexual, demisexual)
Enrollment: 120 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, PhD, Principal Investigator — Yale University
Locations (1):
- Dr. Pachankis' Lab, New York, New York, United States

REFERENCES:
- [Background] Kauer SD, Reid SC, Crooke AH, Khor A, Hearps SJ, Jorm AF, Sanci L, Patton G. Self-monitoring using mobile phones in the early stages of adolescent depression: randomized controlled trial. J Med Internet Res. 2012 Jun 25;14(3):e67. doi: 10.2196/jmir.1858. PMID 22732135
- [Background] Pachankis JE, McConocha EM, Clark KA, Wang K, Behari K, Fetzner BK, Brisbin CD, Scheer JR, Lehavot K. A transdiagnostic minority stress intervention for gender diverse sexual minority women's depression, anxiety, and unhealthy alcohol use: A randomized controlled trial. J Consult Clin Psychol. 2020 Jul;88(7):613-630. doi: 10.1037/ccp0000508. Epub 2020 May 21. PMID 32437174
- [Background] Pachankis JE, Hatzenbuehler ML, Rendina HJ, Safren SA, Parsons JT. LGB-affirmative cognitive-behavioral therapy for young adult gay and bisexual men: A randomized controlled trial of a transdiagnostic minority stress approach. J Consult Clin Psychol. 2015 Oct;83(5):875-89. doi: 10.1037/ccp0000037. Epub 2015 Jul 6. PMID 26147563
- [Result] van Spijker BA, Batterham PJ, Calear AL, Farrer L, Christensen H, Reynolds J, Kerkhof AJ. The suicidal ideation attributes scale (SIDAS): Community-based validation study of a new scale for the measurement of suicidal ideation. Suicide Life Threat Behav. 2014 Aug;44(4):408-19. doi: 10.1111/sltb.12084. Epub 2014 Feb 24. PMID 24612048
- [Result] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Result] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Result] Norman SB, Cissell SH, Means-Christensen AJ, Stein MB. Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety. 2006;23(4):245-9. doi: 10.1002/da.20182. PMID 16688739
- [Result] Radloff, L. S. (1977). The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1(3), 385-401.
- [Result] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in May 2020 and ended in May 2021. Participants for this study were recruited from social media, mobile dating apps, LGBTQ community organizations, and via peer recruitment and referral.
Period: Overall Study
Arm/Group | Online EQuIP | Self-Monitoring
Started | 60 | 60
Baseline | 60 | 60
4-month Post-baseline | 41 | 53
8-month Post-baseline | 48 | 49
Completed | 48 | 49
Not Completed | 12 | 11
Not completed — Lost to Follow-up | 6 | 9
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Dismissal due to ineligibility | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online EQuIP | Self-Monitoring | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.83 (3.00) | 22.03 (3.51) | 21.93 (3.25)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants were asked to select one option for gender identity, with the option to select "other" and indicate their gender identity using a text box.
  Participants
    Gender identity: Cisgender woman | 22 | 29 | 51
    Gender identity: Cisgender man | 10 | 5 | 15
    Gender identity: Transgender woman | 3 | 2 | 5
    Gender identity: Transgender man | 3 | 8 | 11
    Gender identity: Nonbinary (e.g., genderqueer, agender, gender fluid) | 17 | 12 | 29
    Gender identity: Other | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 49 | 49 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were asked to select one option for race/ethnicity, with the option to select "other" and indicate their race/ethnicity using a text box.
  Participants
    Race/ethnicity: American Indian or Alaskan Native | 0 | 1 | 1
    Race/ethnicity: Asian | 12 | 8 | 20
    Race/ethnicity: Black/African American | 1 | 2 | 3
    Race/ethnicity: Native Hawaiian/Pacific Islander | 0 | 0 | 0
    Race/ethnicity: White, Hispanic/Latinx | 6 | 7 | 13
    Race/ethnicity: White, Non-Hispanic/Latinx | 29 | 30 | 59
    Race/ethnicity: Multiracial/Multiple Races | 9 | 11 | 20
    Race/ethnicity: Other | 3 | 1 | 4
Sexual Orientation [Count of Participants; unit: Participants] — Participants were asked to select one option for sexual orientation, with the option to select "other" and indicate their sexual orientation using a text box.
  Participants
    Asexual | 3 | 3 | 6
    Bisexual | 21 | 20 | 41
    Gay | 11 | 8 | 19
    Lesbian | 6 | 14 | 20
    Pansexual | 4 | 4 | 8
    Queer | 11 | 10 | 21
    Other | 4 | 1 | 5
Sex Assigned at Birth [Count of Participants; unit: Participants]
  Female | 42 | 49 | 91
  Male | 17 | 10 | 27
  Intersex | 1 | 1 | 2
Education Degree [Count of Participants; unit: Participants]
  Less than high school | 1 | 1 | 2
  Some high school | 9 | 12 | 21
  High school diploma or GED | 4 | 9 | 13
  Some college | 24 | 17 | 41
  Associate's degree | 1 | 2 | 3
  4-year college degree | 16 | 16 | 32
  Some graduate school | 4 | 2 | 6
  Advanced graduate school degree | 1 | 1 | 2
U.S. Region [Count of Participants; unit: Participants] — U.S. regions were grouped according to U.S. Census Bureau divisions.
  Participants
    Midwest | 11 | 10 | 21
    Northeast | 9 | 13 | 22
    South | 28 | 25 | 53
    West | 12 | 12 | 24
Difficulty Meeting Basic Needs [Count of Participants; unit: Participants] — Participants were asked "How hard is it for you to pay for the very basics, like food, housing, medical care, and utilities now?"
  Participants
    Not very hard | 32 | 33 | 65
    Somewhat hard | 26 | 18 | 44
    Very hard | 2 | 9 | 11
Financial Worry [Mean (Standard Deviation); unit: score on a scale] — Financial worry was assessed by asking participants to rate "How do you feel about your current financial situation?" on a five-point scale (1 = never worry about it; 5 = always worry about it).
  score on a scale | 3.23 (1.01) | 3.23 (1.17) | 3.23 (1.09)

OUTCOME MEASURES:

1. Primary Outcome: Change in Distress
Description: Distress will be measured using the Brief Symptom Inventory (BSI). The BSI is an 18 item measure that uses a 0-4 rating scale for each item. An overall score of 72 would be the highest possible score on the measure and would indicate an extreme level of overall distress.
Time Frame: Baseline, 4 months, 8 months
Population: The decrease in participants from baseline to post-baseline assessments reflect withdrawals, participants lost to follow-up, and participants dismissed from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Online EQuIP | Self-Monitoring
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 1.43 (0.07) | 1.57 (0.09)
  4-month Post-baseline: number analyzed (Participants) | 41 | 53
  4-month Post-baseline | 1.22 (0.11) | 1.34 (0.11)
  8-month Post-baseline: number analyzed (Participants) | 48 | 49
  8-month Post-baseline | 1.07 (0.10) | 1.21 (0.09)

2. Primary Outcome: Change in Depression
Description: Depression will be measured using the Center for Epidemiological Studies -- Depression Scale (CESD). This 20-item measure uses a 0-3 rating (Rarely or none of the time - Most or all of the time) scale and sums across the items with items 3, 11, 14, and 16 reversed. for a minimum score of 0 and a maximum score of 60. Higher scores indicate greater severity of depression. In cases with internally missing data (items not answered), the sums are computed after imputation of the missing values: # items on scale / # actually answered, multiplied by the sum obtained from the answered items. A higher score indicates more depressive symptomatology during the past week.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Online EQuIP | Self-Monitoring
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 14.17 (0.36) | 15.41 (0.47)
  4-month post-baseline: number analyzed (Participants) | 41 | 53
  4-month post-baseline | 12.68 (0.57) | 13.45 (0.50)
  8-month post-baseline: number analyzed (Participants) | 48 | 49
  8-month post-baseline | 12.44 (0.48) | 13.38 (0.50)

3. Primary Outcome: Change in Depression Severity
Description: Depression severity will be measured using the Overall Depression Severity & Impairment Scale (ODSIS). This 5 item measure uses a 0-4 rating scale and sums across the items for a maximum score of 20. The higher the score, the greater the severity of depression.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Online EQuIP | Self-Monitoring
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 7.20 (0.54) | 8.40 (0.58)
  4-month post-baseline: number analyzed (Participants) | 41 | 53
  4-month post-baseline | 6.07 (0.73) | 6.98 (0.58)
  8-month post-baseline: number analyzed (Participants) | 48 | 49
  8-month post-baseline | 6.15 (0.74) | 6.63 (0.73)

4. Primary Outcome: Change in Anxiety Symptoms
Description: Anxiety symptoms will be measured by the Overall Anxiety Severity & Impairment Scale (OASIS). This 5 item measure uses a 0-4 rating scale and sums across the items for a maximum score of 20. The higher the score, the greater the presence of anxiety symptoms.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Online EQuIP | Self-Monitoring
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 9.12 (0.39) | 8.97 (0.44)
  4-month post-baseline: number analyzed (Participants) | 41 | 53
  4-month post-baseline | 7.32 (0.53) | 7.45 (0.51)
  8-month post-baseline: number analyzed (Participants) | 48 | 49
  8-month post-baseline | 7.25 (0.52) | 7.52 (0.60)

5. Primary Outcome: Number of Participants Reporting Any Alcohol Use
Description: Alcohol use in participants will be assessed using the Alcohol Use Disorders Identification (AUDIT) instrument. Any alcohol use over the past 3 months will be measured through the first item of the instrument ("How often, during the last 3 months did you have a drink containing alcohol?") with the creation of a binary variable (1 = any alcohol use, 0 = no alcohol use).
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Online EQuIP | Self-Monitoring
Number analyzed (Participants) | 60 | 60
Participants
  Baseline | 42 | 41
  4-month post-baseline: number analyzed (Participants) | 41 | 53
  4-month post-baseline | 28 | 36
  8-month post-baseline: number analyzed (Participants) | 48 | 49
  8-month post-baseline | 34 | 34

6. Primary Outcome: Number of Participants Reporting Any Suicidal Ideation
Description: Suicidal ideation will be measured using the Suicidal Ideation Attributes Scale (SIDAS). Any suicidal ideation was assessed through the first item of this scale ("In the past month, how often have you had thoughts about suicide?") with the creation of a binary variable (1 = any suicidal ideation, 0 = no suicidal ideation).
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Online EQuIP | Self-Monitoring
Number analyzed (Participants) | 60 | 60
Participants
  Baseline | 37 | 35
  4-month post-baseline: number analyzed (Participants) | 41 | 53
  4-month post-baseline | 25 | 24
  8-month post-baseline: number analyzed (Participants) | 48 | 49
  8-month post-baseline | 28 | 25

7. Primary Outcome: Number of Participants Reporting Any Sexual Risk Behavior
Description: Sexual risk behavior is defined as: condomless anal or vaginal/frontal sex [not counting the sole use of prosthetics] in the absence of PrEP, with any HIV+ partner [except primary HIV+ partners with a known undetectable viral load] or status-unknown partner. A binary variable of any sexual risk behavior was constructed from reports of past-90 day sexual behavior (1 = any sexual risk behavior, 0 = no sexual risk behavior).
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Online EQuIP | Self-Monitoring
Number analyzed (Participants) | 60 | 60
Participants
  Baseline | 4 | 3
  4-month post-baseline: number analyzed (Participants) | 41 | 53
  4-month post-baseline | 2 | 4
  8-month post-baseline: number analyzed (Participants) | 48 | 49
  8-month post-baseline | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline through completion of the final follow-up assessment at 8 months.
Arm/Group | Online EQuIP | Self-Monitoring
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/60
Other Adverse Events (participants affected / at risk) | 1/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Online EQuIP (N=60) | Self-Monitoring (N=60)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Online EQuIP (N=60) | Self-Monitoring (N=60)
Active Suicidality (Psychiatric disorders) | 1 (1) | 0 (0) — Determined by clinician assessment following reports of suicidal ideation as measured by the SIDAS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04408469/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT04408469/SAP_001.pdf